CLINICAL TRIAL: NCT02075372
Title: REgistry of CrossBoss and Hybrid Procedures in FrAnce, the NetheRlands, BelGium and UnitEd Kingdom
Brief Title: CrossBoss and Hybrid Registry on Coronary Chronic Total Occlusions
Acronym: RECHARGE
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Jo Dens, prof. dr., Hasselt University
Other Study IDs: 13/094L
Record Dates: First submitted 2013-12-16; First posted 2014-03-03 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: Chronic Total Occlusion of Coronary Artery; Percutaneous Coronary Intervention; Hybrid; Angioplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data registration of CTO-PCI patients: Patients diagnosed with the presence of one or more chronic total occlusions (CTOs) and who will receive treatment via percutaneous coronary intervention (PCI), which is standard medical practice for these types of lesions. This study will register data on the patients' demographics, CTO characteristics, procedure and outcome. This will be done in the form of a registry.
  Interventions: Other: Data registration

INTERVENTIONS:
Other: Data registration — Patients diagnosed with the presence of one or more chronic total occlusions (CTOs) and who will receive treatment via percutaneous coronary intervention (PCI), which is standard medical practice for these types of lesions. This study will collect data on the patients' demographics, CTO characteristics, procedure and outcome. This will be done in the form of a registry

SUMMARY:
The successful re-opening of a blocked coronary artery has a beneficial effect on the further clinical course (e.g. improvement of clinical symptoms, improved quality of life, increased heart function, etc.). However, some types of blockages are more difficult to open by means of percutaneous coronary intervention (PCI), a procedure which is commonly used for these kind of problems. This procedure makes use of a technique in which special wires, balloons, stents (metal or polymeric tube-like structures) and devices are utilized to re-open or revascularize a blockage in one of the blood vessels of the heart. This type of blockages are chronic total occlusions (CTO). CTOs have certain characteristics which impede the revascularization of the blood vessel.

Nevertheless, remarkable progress has been achieved over the past few years in the area of CTO revascularization or CTO PCI. A large range of CTO dedicated materials, such as guidewires, guiding catheters, devices, balloons and stents, as well as different techniques have been developed. However, at present, reluctance to open CTOs still exists, due to the indications and outcomes of percutaneous revascularization as well as the technical difficulties which commonly arise during these interventional procedures. The presence of these difficulties results in suboptimal success rates worldwide (±70-80%), despite these many innovations.

To increase these success rates and to make sure more interventional cardiologists will treat CTOs, a hybrid treatment algorithm has been developed with the materials (e.g. CrossBoss™ catheter; Bridgepoint Medical, Inc.) and techniques, currently already available. The main purpose of this study is to evaluate the efficacy and efficiency of this hybrid algorithm as well as validating the efficacy of one of the materials (CrossBoss™ catheter), used in this algorithm. To be able to do this, data concerning the patients' demographics, CTO characteristics, procedure and outcome will be collected in the form of a registry. This registry will be performed in several European centra (Belgium, the Netherlands, United Kingdom, France). Since the study will only collect data and no intervention is performed, this will be an observational study. At regular time points, the data will be checked for errors or inconsistencies. To do this, site visits will be performed at pre-defined times.

ELIGIBILITY:
Inclusion Criteria:

* Subject shows the presence of at least one coronary chronic total occlusion (CTO), either with or without the presence of one or more other diseased coronary arteries. This CTO must be located in a native coronary artery and have a visually estimated stenosis of 100%, corresponding with Thrombolysis in Myocardial Infarction (TIMI) flow 0. Following the operators judgment, this occlusion is present for more then 3 months.
* Subject will be/is treated percutaneously for one or more CTOs via the hybrid techniques.
* Subject (or legal guardian) understands the study requirements and the treatment procedures and provides written informed consent before any study-specific procedures are performed.
* Subject is willing to comply with all protocol-required follow-up evaluation (patient will be followed during 1 month after PCI procedure to assess any complications and clinical status).

Exclusion Criteria:

* The occlusion is considered to be less than 3 months present.
* Subject is treated via PCI without application of the hybrid algorithm and/or use of the CrossBoss™ and Stingray™ technology (Bridgepoint Medical, Inc.).
* Subject is participating in another investigational clinical trial that may cause non-compliance with the protocol or confound data interpretation.
* Subject intends to participate in another investigational clinical trial that may cause non-compliance with the protocol or confound data interpretation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with the presence of one or more chronic total occlusions (CTOs) and who will receive treatment via percutaneous coronary intervention (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 1177 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Outcome of CTO PCI procedure | after 3 hours
  Description: Success percentage of the hybrid algorithm and of those procedures in which CrossBoss™ and Stingray™ technologies are used (as a stand alone device or combined with other techniques) in CTO lesions according to the Japanese scoring system (J-CTO). Success is defined as successful revascularization, resulting in TIMI flow 3.

SECONDARY OUTCOMES:
Outcome of PCI procedures in which CrossBoss™ technology is used (as a stand alone device) | after 3 hours
  Outcome (success/failure) of PCI procedures in which CrossBoss™ technology is used (as a stand alone device).
Outcome of PCI procedures in which CrossBoss™ technology is used (combined with other techniques). | after 3 hours
  Outcome (success/failure) of PCI procedures in which CrossBoss™ technology is used (combined with other techniques)
Complications | up to month 1
  Complications (either CrossBoss™/Stingray™ related or not): Major Adverse Cardiac Events (MACE) during in-hospital stay (approximately 1-2 days) and at follow-up (first month after CTO PCI). MACE is common endpoint for death, Q-wave myocardial infarction (MI) (according to ESC guidelines), non Q-wave MI (according to ESC guidelines) and target vessel revascularization. Other complications include target vessel failure (i.e. applies when target vessel is occluded at follow-up (first month after CTO PCI) but no revascularization has been considered), tamponade, perforation, bleeding requiring transfusion/surgery, peri-procedural infarction ((N-)STEMI) (according to ESC guidelines) and loss of side-branches.
Clinical status after PCI procedure | up to month 1
  Record medical drug prescription (after CTO PCI) and clinical status during in-hospital stay and during follow-up (1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Jo Dens, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg; Joren Maeremans, MSc, Study Chair — Ziekenhuis Oost-Limburg
Locations (21):
- Belgium (3):
  - UZ Brussel, Brussels, Limburg
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Hasselt University, Hasselt, Limburg
- France (4):
  - Groupe Hospitalier Mutualiste (GHM), Grenoble
  - Clinique de Marignane, Marignane
  - Nouvelles Cliniques Nantaises (NCN), Nantes
  - Hôpital Nord - CHU de St Etienne, Saint-Priest-en-Jarez
- Netherlands (4):
  - Onze-Lieve-Vrouwe Gasthuis (OLVG), Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht (UMCU), Utrecht
- United Kingdom (10):
  - Basildon University Hospital, Basildon
  - Belfast City Hospital, Belfast
  - University Hospital of Bristol, Bristol
  - Ninewells Hospital, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Golden Jubilee Hospital, Glasgow
  - London Chest Hospital, London
  - Kings College London, London
  - Freeman Hospital, Newcastle
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maeremans J, Dens J, Spratt JC, Bagnall AJ, Stuijfzand W, Nap A, Agostoni P, Wilson W, Hanratty CG, Wilson S, Faurie B, Avran A, Bressollette E, Egred M, Knaapen P, Walsh S; RECHARGE Investigators. Antegrade Dissection and Reentry as Part of the Hybrid Chronic Total Occlusion Revascularization Strategy: A Subanalysis of the RECHARGE Registry (Registry of CrossBoss and Hybrid Procedures in France, the Netherlands, Belgium and United Kingdom). Circ Cardiovasc Interv. 2017 Jun;10(6):e004791. doi: 10.1161/CIRCINTERVENTIONS.116.004791. PMID 28625964